CLINICAL TRIAL: NCT04775875
Title: Open Label Study for the Use of Transcranial Ultrasound Treatment of Obsessive-Compulsive Disorder
Brief Title: The Use of Transcranial Ultrasound Treatment of Obsessive-Compulsive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fUS-OCD
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Active (Experimental): Patients will undergo ten to thirty minutes of transcranial ultrasound treatment. The sonification device will be aimed at the caudate. Targeting will include reference to scalp fiducials based on the obtained MRI; confirmation of target accuracy will either be obtained by Doppler waveform confirmation or optical tracking technology which co-registers patient neuroimaging with real space.
  Interventions: Device: Focused Ultrasound

INTERVENTIONS:
Device: Focused Ultrasound — The DWL Doppler ultrasound device enables visual and auditory wave form confirmation of cerebral arteries, and optical tracking technology (eg, AntNeuro Visor2 system) may be used in tandem with the Brainsonix Pulsar 1002 ultrasound device to track a patient's brain in virtual space as well as their physical location, thereby ensuring accurate placement.
  Other Names: Brainsonix; DWL

SUMMARY:
The primary objective of this study is to determine the safety and efficacy of ultrasound as a treatment for Obsessive Compulsive disorder.

DETAILED DESCRIPTION:
The present study is being undertaken as an open-label study to evaluate the safety and feasibility of focused ultrasound as an intervention for patients with obsessive compulsive disorder (OCD). Participants in this study will undergo 8 consecutive weekly sessions of transcranial low-intensity focused ultrasound (LIFUP) targeting the caudate of the basal ganglia. The safety of this protocol will be closely monitored and data will be used to determine whether any significant safety issues exist when using focused ultrasound for this neurological application. Treatment response will be measured using the Beck Depression & Anxiety Inventories, the Yale-Brown Obsessive-Compulsive Scale, and the Global Rating of Change Scale.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Obsessive Compulsive Disorder
* Score greater than 15 on the Yale-Brown Obsessive Compulsive Scale (Y- BOCS)
* Failure to remit with 3 SSRIs, antidepressants and/or anxiolytics
* Must be willing to comply with the study protocol
* English Proficiency
* At least 18 years of age

Exclusion Criteria:

* Subjects not English proficient
* Subjects unable to give informed con-sent
* Subjects who would not be able to lay down without excessive movement in a calm environment sufficiently long enough to be able to achieve sleep
* Pregnancy, women who may become pregnant or are breastfeeding
* Advanced terminal illness
* Any active cancer or chemotherapy
* Any other neoplastic illness or illness characterized by neovascularity
* Macular degeneration
* Subjects with scalp rash or open wounds on the scalp (for example from treatment of squamous cell cancer)
* Advanced kidney, pulmonary, cardiac or liver failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Disorder Scale (Y-BOC) | Baseline
  This instrument is designed to evaluate the severity of symptoms for Obsessive Compulsive Disorder. The Y-BOC is composed of 10 items, and uses a scale that ranges from 0-4 based on the individuals mark going from 0 as no symptoms to 4 extreme symptoms for a total possible score of 40. Severity range is as follows: subclinical OCD is indicated by scores ranging from 0-7, mild OCD is indicated by scores ranging from 8-15, moderate OCD is indicated by scores ranging from 16-23, severe OCD is indicated by scores ranging from 24-31, and extreme OCS is indicated by scores ranging from 32-40. Moderate to extreme symptoms are clinically significant. For treatment of OCD, a clinically significant change must decrease greater than or equal to 35% relative to baseline. This amount of change is also most predictive of treatment response.
Beck Anxiety Inventory (BAI) | Baseline
  The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety symptoms. Each of the 21 items asks whether the patient has experienced various anxiety symptoms in the last two weeks, and if so, how severely. Each question/answer is scored on a scale value of "0" (not at all) to "3" (severely). Higher total scores indicate more severe anxiety symptoms. The maximum total score possible is 63 points. The standard cutoff scores are: 0-7 = minimal anxiety; 8-15 = mild anxiety; 16-25 = moderate anxiety; 26-63 = severe anxiety. A reduction in score by at least 30% is considered clinically meaningful.
Beck Depression Inventory (BDI-II) | Baseline
  The BDI-II is a 21-question multiple-choice self-report inventory. Each question involves four possible responses, ranging in intensity from "0" (this item does not apply) to "3" (this item applies severely). The test is scored as the sum of all of the response values; this number is used to determine the severity of depressive symptoms. A score of 0 to 3 is possible for each question with a maximum total score of 63 points. The standard cutoff scores are as follows: 0-13 total points = minimal depression; 14-19 total points = mild depression; 20-28 total points = moderate depression; and 29-63 total points = severe depression. A reduction in the total score by at least 30% is considered to be clinically significant.
Global Rating of Change (GRC) | Baseline
  The GRC consists of a single likert-scale ranging from "-5" (very much worse) to "0" (neutral/no change) to "5" (very much better). The GRC is obtained in an interview format to assess a patient's perceived change in status following a treatment. A score that is at least 2 or greater is considered to indicate clinically significant change.

SECONDARY OUTCOMES:
Yale-Brown Obsessive Compulsive Disorder Scale (Y-BOC) | 8 weeks from baseline
  This instrument is designed to evaluate the severity of symptoms for Obsessive Compulsive Disorder. The Y-BOC is composed of 10 items, and uses a scale that ranges from 0-4 based on the individuals mark going from 0 as no symptoms to 4 extreme symptoms for a total possible score of 40. Severity range is as follows: subclinical OCD is indicated by scores ranging from 0-7, mild OCD is indicated by scores ranging from 8-15, moderate OCD is indicated by scores ranging from 16-23, severe OCD is indicated by scores ranging from 24-31, and extreme OCS is indicated by scores ranging from 32-40. Moderate to extreme symptoms are clinically significant. For treatment of OCD, a clinically significant change must decrease greater than or equal to 35% relative to baseline. This amount of change is also most predictive of treatment response.
Beck Anxiety Inventory (BAI) | 8 weeks from baseline
  The BAI is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety symptoms. Each of the 21 items asks whether the patient has experienced various anxiety symptoms in the last two weeks, and if so, how severely. Each question/answer is scored on a scale value of "0" (not at all) to "3" (severely). Higher total scores indicate more severe anxiety symptoms. The maximum total score possible is 63 points. The standard cutoff scores are: 0-7 = minimal anxiety; 8-15 = mild anxiety; 16-25 = moderate anxiety; 26-63 = severe anxiety. A reduction in score by at least 30% is considered clinically meaningful.
Beck Depression Inventory (BDI-II) | 8 weeks from baseline
  The BDI-II is a 21-question multiple-choice self-report inventory. Each question involves four possible responses, ranging in intensity from "0" (this item does not apply) to "3" (this item applies severely). The test is scored as the sum of all of the response values; this number is used to determine the severity of depressive symptoms. A score of 0 to 3 is possible for each question with a maximum total score of 63 points. The standard cutoff scores are as follows: 0-13 total points = minimal depression; 14-19 total points = mild depression; 20-28 total points = moderate depression; and 29-63 total points = severe depression. A reduction in the total score by at least 30% is considered to be clinically significant.
Global Rating of Change (GRC) | 8 weeks from baseline
  The GRC consists of a single likert-scale ranging from "-5" (very much worse) to "0" (neutral/no change) to "5" (very much better). The GRC is obtained in an interview format to assess a patient's perceived change in status following a treatment. A score that is at least 2 or greater is considered to indicate clinically significant change.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, MD, Principal Investigator — Neurological Associates of West LA
Locations (2):
- United States (2):
  - Neurological Associates of West LA, Santa Monica, California
  - Neurological Associates of West Los Angeles, Santa Monica, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bloch MH, Landeros-Weisenberger A, Kelmendi B, Coric V, Bracken MB, Leckman JF. A systematic review: antipsychotic augmentation with treatment refractory obsessive-compulsive disorder. Mol Psychiatry. 2006 Jul;11(7):622-32. doi: 10.1038/sj.mp.4001823. Epub 2006 Apr 4. PMID 16585942
- [Background] Rapoport JL. Obsessive compulsive disorder and basal ganglia dysfunction. Psychol Med. 1990 Aug;20(3):465-9. doi: 10.1017/s0033291700016962. No abstract available. PMID 2236357
- [Background] Welter ML, Burbaud P, Fernandez-Vidal S, Bardinet E, Coste J, Piallat B, Borg M, Besnard S, Sauleau P, Devaux B, Pidoux B, Chaynes P, Tezenas du Montcel S, Bastian A, Langbour N, Teillant A, Haynes W, Yelnik J, Karachi C, Mallet L; French Stimulation dans Trouble Obsessionnel Compulsif (STOC) Study Group. Basal ganglia dysfunction in OCD: subthalamic neuronal activity correlates with symptoms severity and predicts high-frequency stimulation efficacy. Transl Psychiatry. 2011 May 3;1(5):e5. doi: 10.1038/tp.2011.5. PMID 22832400